CLINICAL TRIAL: NCT01493557
Title: A Prospective, Open Label Study Evaluating the Efficacy of Two Management Strategies (Pantoprazole 40 mg q.a.m. and Taking Pradaxa® With Food (Within 30 Minutes After a Meal) on Gastrointestinal Symptoms (GIS) in Patients Newly on Treatment With Pradaxa® 150 mg b.i.d., 110 mg b.i.d. or 75 mg b.i.d. for the Prevention of Stroke and Systemic Embolism in Patients With Non-valvular Atrial Fibrillation (NVAF)
Brief Title: A Prospective, Open Label Study Evaluating Two Management Strategies on Gastrointestinal Symptoms in Patients Newly on Treatment With Pradaxa for the Prevention of Stroke and Systemic Embolism With Non-valvular Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1160.128
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Pantoprazole; Dabigatran; Postprandial Period

ARMS (3):
- Pradaxa (dabigaran etexilate) (Other): Patients with non valvular atrial fibrillation for whom Pradaxa is indicated in accordance with the current local label, not previously treated with Pradaxa, will be provided 3 months of treatment for the prevention of stroke and systemic embolism. Patients who report gastrointestinal symptoms (GIS) will be randomized to one of two management strategies, and data documenting the intensity and duration of the GIS will be collected.
  Interventions: Drug: Pradaxa (dabigatran etexilate)
- Pradaxa and pantoprazole (Active Comparator): Patients that develop gastrointestinal symptoms (GIS) will be randomized 1:1 to either pantoprazole 40 mg q.a.m., p.o., or taking Pradaxa (dabigatran etexilate) within 30 minutes after a meal
  Interventions: Drug: pantoprazole; Drug: Pradaxa (dabigatran etexilate)
- Pradaxa, 30 minutes after a meal (Active Comparator): Patients that develop gastrointestinal symptoms (GIS) will be randomized 1:1 to either pantoprazole 40 mg q.a.m., p.o., or taking Pradaxa (dabigatran etexilate) within 30 minutes after a meal
  Interventions: Drug: Pradaxa, within 30 minutes after a meal

INTERVENTIONS:
Drug: pantoprazole — 40 mg q.a.m, p.o.
  Arms: Pradaxa and pantoprazole
Drug: Pradaxa (dabigatran etexilate) — 150 mg or 75 mg b.i.d. (150 mg or 110 mg b.i.d. in Canada)
  Arms: Pradaxa (dabigaran etexilate)
Drug: Pradaxa, within 30 minutes after a meal — Patients randomized to this intervention would be instructed to take their dabigatran 30 minutes after a meal
  Arms: Pradaxa, 30 minutes after a meal
Drug: Pradaxa (dabigatran etexilate) — 150 mg or 75 mg b.i.d. (150 mg or 110 mg b.i.d. in Canada)
  Arms: Pradaxa and pantoprazole

SUMMARY:
This is a prospective and open label study that aims to enroll approximately 1200 patients with non-valvular atrial fibrillation (NVAF) not previously treated with Pradaxa® and free of gastrointestinal symptoms (GIS) for at least 2 weeks prior to enrolment. Approximately 125 sites in North America will be recruited. Patients who report GIS during the 3 month treatment period will be randomized to one of two management strategies, and data documenting the intensity and duration of the GIS will be collected.

ELIGIBILITY:
Inclusion criteria:

1. Documented non-valvular atrial fibrillation (NVAF) for whom Pradaxa® (dabigatran etexilate) is indicated per the current local label, but who have not received treatment with Pradaxa® (dabigatran etexilate), or who have not been started on Pradaxa® (dabigatran etexilate) more than 7 days prior to potential enrolment in the study. NVAF may be documented by 12-lead electrocardiogram, rhythm strip, pacemaker/ implantable cardioverter defibrillator (ICD) electrograms or Holter monitoring
2. Male and female patients, age greater than or equal to 18 years at entry
3. Written, informed consent

Exclusion criteria:

1. History within 2 weeks of any of the following gastrointestinal (GI) disorders: heartburn, indigestion, gastritis, upper abdominal pain or discomfort, or gastroesophageal reflux requiring the use of proton pump inhibitors, histamine-2 receptor blockers or antacids. Patients with nausea and/or vomiting within the 2 weeks are not excluded if the symptoms were clearly associated with a self-limited acute or febrile illness. Short-term use of PPIs, as prophylaxis, in a hospital setting for the prevention of stress ulcers is acceptable. Calcium carbonate supplements for calcium replacement is not exclusionary (as long as these products are being used as calcium supplementation/replacement and are not being used to treat or relieve GIS.)
2. GI bleeding within one year or any history of symptomatic or endoscopically documented gastroduodenal ulcer or diverticulitis, unless the cause has been permanently eliminated by medical therapy or by surgery(e.g., patients with peptic ulcer disease with endoscopically proven cure after therapy or lower GI bleeding due to diverticulosis cured by segmental colectomy are not excluded.)
3. not applicable
4. Contraindication to pantoprazole or other proton pump inhibitors, e.g. omeprazole, lansoprazole, rabeprazole, atnoprazole, esomeprazole
5. Contraindication to Pradaxa® (dabigatran etexilate) or known hypersensitivity to Pradaxa® (dabigatran etexilate) or its excipients
6. Hemorrhagic disorder, bleeding diathesis or active pathological bleeding
7. Need for anticoagulant treatment for disorders other than atrial fibrillation
8. Current treatment with rifampin
9. Creatinine clearance <15ml/min (in Canada, <30ml/min), or patients on renal replacement therapy (dialysis)
10. Pre-menopausal women (last menstruation less than or equal to 1 year prior to informed consent) who: are nursing or pregnant, or are of child bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study. Acceptable methods of birth control include abstinence, tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral implantable or injectable contraceptives, double barrier method and vasectomized partner.
11. Patients who have received an investigational drug in the past 30 days or are participating in another drug study
12. Patients considered unreliable by the investigator concerning the requirements for follow-up during the study
13. Any condition the investigator believes would not allow safe participation in the study
14. Contraindication in patients with mechanical heart valves. The use of Pradaxa in the setting of other forms of valvular heart disease, including the presence of a bio-prosthetic valve, is not recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (103):
- United States (81):
  - 1160.128.1046 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.128.1045 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1160.128.1003 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1160.128.1093 Boehringer Ingelheim Investigational Site, Chandler, Arizona
  - 1160.128.1067 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1160.128.1103 Boehringer Ingelheim Investigational Site, Mesa, California
  - 1160.128.1094 Boehringer Ingelheim Investigational Site, Newport Beach, California
  - 1160.128.1042 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.128.1005 Boehringer Ingelheim Investigational Site, Colorado Spring, Colorado
  - 1160.128.1023 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1160.128.1016 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.128.1066 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.128.1018 Boehringer Ingelheim Investigational Site, Guilford, Connecticut
  - 1160.128.1050 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1160.128.1057 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1160.128.1085 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1160.128.1111 Boehringer Ingelheim Investigational Site, Atlantis, Florida
  - 1160.128.1032 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 1160.128.1021 Boehringer Ingelheim Investigational Site, Coral Springs, Florida
  - 1160.128.1027 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 1160.128.1019 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.128.1062 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.128.1054 Boehringer Ingelheim Investigational Site, Largo, Florida
  - 1160.128.1097 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1160.128.1109 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1160.128.1087 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1160.128.1058 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.128.1007 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.128.1060 Boehringer Ingelheim Investigational Site, Rockledge, Florida
  - 1160.128.1096 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1160.128.1068 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1160.128.1076 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1160.128.1073 Boehringer Ingelheim Investigational Site, Melrose Park, Illinois
  - 1160.128.1048 Boehringer Ingelheim Investigational Site, Winfield, Illinois
  - 1160.128.1105 Boehringer Ingelheim Investigational Site, Hammond, Indiana
  - 1160.128.1029 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.128.1079 Boehringer Ingelheim Investigational Site, Overland Park, Kansas
  - 1160.128.1008 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1160.128.1025 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1160.128.1100 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 1160.128.1041 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1160.128.1012 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.128.1015 Boehringer Ingelheim Investigational Site, Rochester Hills, Michigan
  - 1160.128.1004 Boehringer Ingelheim Investigational Site, Tupelo, Mississippi
  - 1160.128.1014 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 1160.128.1047 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1160.128.1075 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.128.1069 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 1160.128.1011 Boehringer Ingelheim Investigational Site, Kalispell, Montana
  - 1160.128.1092 Boehringer Ingelheim Investigational Site, Lincoln, Nebraska
  - 1160.128.1059 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1160.128.1039 Boehringer Ingelheim Investigational Site, Elmer, New Jersey
  - 1160.128.1035 Boehringer Ingelheim Investigational Site, Flemington, New Jersey
  - 1160.128.1036 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1160.128.1063 Boehringer Ingelheim Investigational Site, Hawthorne, New York
  - 1160.128.1078 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1160.128.1001 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 1160.128.1022 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1160.128.1052 Boehringer Ingelheim Investigational Site, Gastonia, North Carolina
  - 1160.128.1071 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1160.128.1091 Boehringer Ingelheim Investigational Site, Gallipolis, Ohio
  - 1160.128.1107 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1160.128.1053 Boehringer Ingelheim Investigational Site, Bend, Oregon
  - 1160.128.1033 Boehringer Ingelheim Investigational Site, Hillsboro, Oregon
  - 1160.128.1037 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1160.128.1034 Boehringer Ingelheim Investigational Site, Camp Hill, Pennsylvania
  - 1160.128.1010 Boehringer Ingelheim Investigational Site, Langhorne, Pennsylvania
  - 1160.128.1056 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.128.1065 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1160.128.1043 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1160.128.1040 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 1160.128.1006 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1160.128.1104 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1160.128.1061 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1160.128.1090 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 1160.128.1082 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.128.1102 Boehringer Ingelheim Investigational Site, Layton, Utah
  - 1160.128.1077 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 1160.128.1064 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 1160.128.1110 Boehringer Ingelheim Investigational Site, Manassas, Virginia
  - 1160.128.1099 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- Canada (22):
  - 1160.128.1160 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.128.1159 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.128.1152 Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - 1160.128.1153 Boehringer Ingelheim Investigational Site, Spruce Grove, Alberta
  - 1160.128.1167 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1160.128.1158 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.128.1154 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1160.128.1166 Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - 1160.128.1151 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1160.128.1168 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.128.1164 Boehringer Ingelheim Investigational Site, Collingwood, Ontario
  - 1160.128.1173 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1160.128.1171 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1160.128.1156 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.128.1157 Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - 1160.128.1155 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1160.128.1170 Boehringer Ingelheim Investigational Site, Peterborough, Ontario
  - 1160.128.1165 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1160.128.1169 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1160.128.1161 Boehringer Ingelheim Investigational Site, Stayner, Ontario
  - 1160.128.1162 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.128.1172 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] O'Dea D, Whetteckey J, Ting N. A Prospective, Randomized, Open-Label Study to Evaluate Two Management Strategies for Gastrointestinal Symptoms in Patients Newly on Treatment with Dabigatran. Cardiol Ther. 2016 Dec;5(2):187-201. doi: 10.1007/s40119-016-0071-5. Epub 2016 Oct 5. PMID 27709460

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Prospective, randomized, open label trial. 1067 patients treated with Pradaxa and 117 patients were randomized to a management strategy. NVAF= non-valvular atrial fibrillation and GIS = gastrointestinal symptoms.
Groups:
- Pradaxa, 30 Minutes After a Meal (Randomized): Randomized patients that develop gastrointestinal symptoms (GIS) were orally administered to Pradaxa (dabigatran etexilate) 150 mg or Pradaxa (dabigatran etexilate) 75 mg twice daily ( b.i.d.) taken with food (150 mg or 110 mg b.i.d. in Canada), within 30 minutes after a meal (4 weeks).
- Pantoprazole 40 mg (Randomized): Randomized patients that develop gastrointestinal symptoms (GIS) were orally administered to delayed release tablet pantoprazole 40 mg once daily in the Morning (q.a.m) (4 weeks).
- Pradaxa, Never Randomized: Patients who were treated for 3 months with Pradaxa ® and were never randomized to management strategies.
Period: Not Randomized to Management Strategies
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized) | Pradaxa, Never Randomized
Started | 0 | 0 | 950
Without Experiencing GIS | 0 | 0 | 854 (754 patients completed the trial.)
Reported GIS Prior to EOT Visit | 0 | 0 | 48 (32 patients completed the trial.)
Reported GIS Only at EOT Visit | 0 | 0 | 48 (26 patients completed (GIS resolved ) and 4 patients completed (GIS not resolved ) the trial.)
Completed | 0 | 0 | 816
Not Completed | 0 | 0 | 134
Not completed — Worsening of events associate with NVAF. | 0 | 0 | 1
Not completed — Worsening of other pre-existing disease | 0 | 0 | 9
Not completed — Other adverse event | 0 | 0 | 54
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 10
Not completed — Early termination | 0 | 0 | 34
Not completed — Other than stated above | 0 | 0 | 21
Period: Randomized to Management Strategies
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized) | Pradaxa, Never Randomized
Started | 59 | 58 | 0
Completed | 44 | 47 | 0
Not Completed | 15 | 11 | 0
Not completed — Worsening of events associate with GIS | 3 | 2 | 0
Not completed — Other adverse event | 8 | 5 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Other than stated above | 1 | 3 | 0
Period: Adding the Second Strategy
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized) | Pradaxa, Never Randomized
Started | 14 | 15 | 0
Completed | 12 | 11 | 0
Not Completed | 2 | 4 | 0
Not completed — Worsening of events associate with GIS | 1 | 1 | 0
Not completed — Other adverse event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Entered Set (ES): This patient set included all patients entered in the study. For those patients who were randomized to management strategies, their data prior to randomization was included in the entered set. All data from patients who were never randomized are in the entered set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized) | Pradaxa, Never Randomized | Total
Number analyzed (Participants) | 59 | 58 | 950 | 1067
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (11.1) | 69.6 (10.8) | 69.7 (10.7) | 69.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 304 | 346
  Male | 37 | 38 | 646 | 721

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Complete Effectiveness of Initial GIS Management Strategy
Description: The percentage of patients experiencing complete relief of gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) vs. administration of Pradaxa® (dabigatran etexilate) within 30 minutes after a meal at 4 weeks.
  Complete effectiveness is defined as at the time of evaluation, both primary GIS and secondary GIS are all resolved.
Time Frame: Week 4
Population: Full Analysis Set (FAS): This patient set included all patients who developed GIS and who were randomized into the two management strategies.
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants | 55.9 | 67.2
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); Evaluation of GIS was based on Last observation carried forward (LOCF) data up to the last observed time or up to adding the second management strategy; Test type: Superiority or Other; p = 0.2554, Fisher Exact; Mean Difference (Final Values) = 11.31, 95% CI 2-sided [-6.54 to 29.49] — Exact 95% Confidence interval (CI) and the difference between the two strategies were calculated using the Clopper Pearson approach

2. Secondary Outcome: Rate of Partial Effectiveness of Initial GIS Management Strategies
Description: The percentage of patients experiencing partial relief of gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) and patients taking Pradaxa® (dabigatran etexilate) within 30 minutes after a meal at 4 weeks.
  Partial effectiveness is defined as at the time of evaluation, either primary GIS is improved; or primary GIS is resolved, but there were still un-resolved secondary GIS.
Time Frame: Week 4
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants | 11.9 | 19.0
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3165, Fisher Exact; Mean Difference (Final Values) = 7.10, 95% CI 2-sided [-11.24 to 24.58] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Combined Rate of Complete or Partial Effectiveness of Initial GIS Management Strategies
Description: The percentage of patients experiencing complete or partial effectiveness of gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) vs. administration of Pradaxa ® (dabigatran etexilate) within 30 minutes after a meal at 4 weeks.
  Complete effectiveness is defined as at the time of evaluation, both primary GIS and secondary GIS are all resolved. Partial effectiveness is defined as at the time of evaluation, either primary GIS is improved; or primary GIS is resolved, but there were still un-resolved secondary GIS.
Time Frame: Week 4
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants | 67.8 | 86.2
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0273, Fisher Exact; Mean Difference (Final Values) = 18.41, 95% CI 2-sided [0.71 to 35.98] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Rate of Complete Effectiveness of Combined GIS Management Strategies
Description: The percentage of patients experiencing complete relief of combined gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) vs. administration of Pradaxa ® (dabigatran etexilate) within 30 minutes after a meal.
  Complete effectiveness is defined as at the time of evaluation, both primary GIS and secondary GIS are all resolved.
Time Frame: Week 8
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 14 | 15
percentage of participants | 42.9 | 33.3
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7104, Fisher Exact; Mean Difference (Final Values) = -9.52, 95% CI 2-sided [-44.22 to 28.40] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Rate of Partial Effectiveness of Combined GIS Management Strategies
Description: The percentage of patients experiencing partial relief of gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) vs. administration of Pradaxa ® (dabigatran etexilate) within 30 minutes after a meal at 4 weeks.
  Partial effectiveness is defined as at the time of evaluation, either primary GIS is improved; or primary GIS is resolved, but there were still un-resolved secondary GIS.
Time Frame: Week 8
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 14 | 15
percentage of participants | 42.9 | 46.7
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = 3.81, 95% CI 2-sided [-32.94 to 40.44] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Combined Rate of Complete or Partial Effectiveness of Combined GIS Management Strategies
Description: The percentage of patients experiencing combined of complete or partial relief of gastrointestinal symptoms (GIS) when taking pantoprazole 40 mg once daily in the morning (q.a.m.) vs. administration of Pradaxa ® (dabigatran etexilate) within 30 minutes after a meal.
  Complete effectiveness is defined as at the time of evaluation, both primary GIS and secondary GIS are all resolved. Partial effectiveness is defined as at the time of evaluation, either primary GIS is improved; or primary GIS is resolved, but there were still un-resolved secondary GIS.
Time Frame: Week 8
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 14 | 15
percentage of participants | 85.7 | 80.0
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = -5.71, 95% CI 2-sided [-41.25 to 28.77] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Rates of Complete Effectiveness of GIS at Each Visit.
Description: The percentage of patients experiencing complete effectiveness of gastrointestinal symptoms (GIS) at each visit by management strategy.
  Evaluation of GIS was based on Last observation carried forward (LOCF) data up to the last observed time or up to adding the second management strategy.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 & Week 8
Population: Full analysis Set (FAS).
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants
  Baseline (n= 59 , 58) | 0.0 | 0.0
  GIS 3 (Week 1, n= 59 , 58) | 39.0 | 51.7
  GIS 4 (Week 2, n= 59 , 58) | 45.8 | 55.2
  GIS 5 (Week 3, n= 59 , 58) | 55.9 | 60.3
  GIS 6 (Week 4, n= 59 , 58) | 55.9 | 67.2
  GIS 7 (Week 5, n= 14 , 15) | 28.6 | 40.0
  GIS 8 (Week 6, n= 14 , 15) | 42.9 | 40.0
  GIS 9 (Week 7, n= 14 , 15) | 42.9 | 33.3
  GIS 10 (Week 8, n= 14 , 15) | 42.9 | 33.3

8. Secondary Outcome: Rates of Partial Effectiveness of GIS at Each Visit.
Description: The percentage of patients experiencing partial effectiveness of gastrointestinal symptoms (GIS) at each visit by management strategy.
  Evaluation of GIS was based on Last observation carried forward (LOCF) data up to the last observed time or up to adding the second management strategy.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 & Week 8
Population: Full Analysis Set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants
  Baseline (n= 59 , 58) | 0.0 | 0.0
  GIS 3 (Week 1, n= 59 , 58) | 16.9 | 13.8
  GIS 4 (Week 2, n= 59 , 58) | 13.6 | 24.1
  GIS 5 (Week 3, n= 59 , 58) | 8.5 | 22.4
  GIS 6 (Week 4, n= 59 , 58) | 11.9 | 19.0
  GIS 7 (Week 5, n= 14 , 15) | 21.4 | 40.0
  GIS 8 (Week 6, n= 14 , 15) | 42.9 | 40.0
  GIS 9 (Week 7, n= 14 , 15) | 42.9 | 46.7
  GIS 10 (Week 8, n= 14 , 15) | 42.9 | 46.7

9. Secondary Outcome: Rates of Complete or Partial Effectiveness of GIS at Each Visit.
Description: The percentage of patients experiencing complete or partial effectiveness of gastrointestinal symptoms (GIS) at each visit by management strategy.
  Evaluation of GIS was based on Last observation carried forward (LOCF) data up to the last observed time or up to adding the second management strategy.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 & Week 8
Population: Full Analysis Set (FAS).
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
percentage of participants
  Baseline (n= 59 , 58) | 0.0 | 0.0
  GIS 3 (Week 1, n= 59 , 58) | 55.9 | 65.5
  GIS 4 (Week 2, n= 59 , 58) | 59.3 | 79.3
  GIS 5 (Week 3, n= 59 , 58) | 64.4 | 82.8
  GIS 6 (Week 4, n= 59 , 58) | 67.8 | 86.2
  GIS 7 (Week 5, n= 14 , 15) | 50.0 | 80.0
  GIS 8 (Week 6, n= 14 , 15) | 85.7 | 80.0
  GIS 9 (Week 7, n= 14 , 15) | 85.7 | 80.0
  GIS 10 (Week 8, n= 14 , 15) | 85.7 | 80.0

10. Secondary Outcome: Time Between Symptom Onset and First Observed Complete or Partial Effectiveness and Between Symptom Onset and Last Observed Symptom
Description: Time between symptom onset and first observed complete or partial effectiveness and between symptom onset and last observed symptom by management strategy.
Time Frame: Week 8
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized)
Number analyzed (Participants) | 59 | 58
days
  Duration of GIS (N= 58; 58) | 23.5 (25.67) | 23.9 (25.35)
  Time to first complete effectiveness (N= 43; 50) | 12.1 (13.45) | 10.7 (10.23)
  Time to first partial effectiveness(N= 6; 2) | 23.7 (15.50) | 3.5 (2.12)
Statistical Analysis 1: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); Mean difference for the Duration of gastrointestinal symptoms (GIS); Test type: Superiority or Other; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-9.9 to 8.9] — Mean difference = (Mean number of days for Pradaxa w/meal) - (Mean number of days for pantoprazole)
Statistical Analysis 2: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); Mean difference for Time to first complete effectiveness. Complete effectiveness of a gastrointestinal symptoms (GIS) management strategy can only be measured at a point in time. Because the same or a different GIS could occur after a time of effective GIS management, the patients who indicated some degree of effectiveness at one visit may not be the same patients who experience effectiveness at a subsequent visit; Test type: Superiority or Other; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-3.5 to 6.3] — Mean difference = (Mean number of days for Pradaxa w/meal) - (Mean number of days for pantoprazole)
Statistical Analysis 3: Comparison: Pradaxa, 30 Minutes After a Meal (Randomized) vs Pantoprazole 40 mg (Randomized); Mean difference for Time to first complete effectiveness. Partial effectiveness of a gastrointestinal symptoms (GIS) management strategy can only be measured at a point in time. Because the same or a different GIS could occur after a time of effective GIS management, the patients who indicated some degree of effectiveness at one visit may not be the same patients who experience effectiveness at a subsequent visit; Test type: Superiority or Other; Mean Difference (Final Values) = 20.2, 95% CI 2-sided [-8.2 to 48.5] — Mean difference = (Mean number of days for Pradaxa w/meal) - (Mean number of days for pantoprazole)

ADVERSE EVENTS:
Time Frame: From first drug administration until 6 days after end of trial, up to 158 days.
Arm/Group | Pradaxa, 30 Minutes After a Meal (Randomized) | Pantoprazole 40 mg (Randomized) | Pradaxa, Never Randomized
Serious Adverse Events (participants affected / at risk) | 2/59 | 3/58 | 109/950
Other Adverse Events (participants affected / at risk) | 37/59 | 35/58 | 161/950
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pradaxa, 30 Minutes After a Meal (Randomized) (N=59) | Pantoprazole 40 mg (Randomized) (N=58) | Pradaxa, Never Randomized (N=950)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 22
Atrial flutter (Cardiac disorders) | 0 | 0 | 4
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 21
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 3
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Congenital cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Colon dysplasia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 5
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Gangrene (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 5
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 1
Heart rate decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 3
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 5
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pradaxa, 30 Minutes After a Meal (Randomized) (N=59) | Pantoprazole 40 mg (Randomized) (N=58) | Pradaxa, Never Randomized (N=950)
Abdominal discomfort (Gastrointestinal disorders) | 7 | 13 | 25
Abdominal distension (Gastrointestinal disorders) | 8 | 12 | 23
Abdominal pain upper (Gastrointestinal disorders) | 8 | 10 | 26
Constipation (Gastrointestinal disorders) | 3 | 4 | 12
Defaecation urgency (Gastrointestinal disorders) | 4 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 30
Dyspepsia (Gastrointestinal disorders) | 17 | 15 | 73
Epigastric discomfort (Gastrointestinal disorders) | 9 | 10 | 18
Eructation (Gastrointestinal disorders) | 13 | 10 | 25
Faeces hard (Gastrointestinal disorders) | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 5 | 5 | 14
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 10 | 31
Regurgitation (Gastrointestinal disorders) | 9 | 4 | 15
Dizziness (Nervous system disorders) | 3 | 2 | 20
Bronchitis (Infections and infestations) | 3 | 1 | 18
Headache (Nervous system disorders) | 1 | 3 | 11

LIMITATIONS AND CAVEATS:
The modest sample size,non-specific nature of symptoms,&reliance on patient self-reporting of their symptoms may contributed some bias to the final result.An open-label design may lead to patient/investigator bias in reporting symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.